CLINICAL TRIAL: NCT04404920
Title: An Observational Study of the Frequency of Oral Symptoms in Patients With Advanced Cancer
Brief Title: Oral Assessment of Symptoms in Advanced Cancer
Acronym: OASis
Status: Completed | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OASis study
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Oral Complication; Cancer
Keywords: Oral symptoms; Cancer; Palliative care
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Novel questionnaire about oral symptoms ("Oral symptom assessment scale / OSAS), and validated questionnaire about physical and psychological symptoms (Memorial Symptom Assessment Scale / MSAS).

SUMMARY:
Observational study of prevalence of oral symptoms in patients with advanced cancer using a novel questionnaire ("Oral symptom assessment scale")

DETAILED DESCRIPTION:
A novel questionnaire (the "Oral symptom assessment scale" / OSAS) has been developed to assess a range of oral symptoms in patients with advanced cancer.

The OSAS consists of 20 symptoms, which were chosen following a review of the literature / discussion with experts in the field. The OSAS was modelled on the Memorial Symptom Assessment Scale (MSAS), and asks about the presence of the symptoms, the frequency of the symptoms (i.e. "rarely"; "occasionally"; "frequently"; or "almost constantly"), the severity of the symptoms (i.e. "slight"; "moderate"; "severe"; or "very severe"), and how much distress they cause (i.e. "not at all"; "a little bit"; "somewhat"; "quite a bit"; or "very much"). The questions relate to the last week.

Patients will be given the OSAS to complete, and also the short form of the MSAS (which asks about the presence, and related distress, of 32 physical / psychological symptoms, including a small number of oral symptoms). Demographic data, cancer diagnosis, and performance status will also be collected. The study involves a single visit / assessment.

Descriptive statistics will be used to present the data, and hierarchical cluster analysis will be used to identify oral symptom clusters. Kappa tests will be used to compare analogous questions on the OSAS and short form MSAS (as part of the validation of the OSAS).

ELIGIBILITY:
Inclusion Criteria:

* age > 18yr; diagnosis of locally advanced / metastatic cancer; already known to the specialist palliative care team

Exclusion Criteria:

* inability to give informed consent; inability to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 subjects that are either inpatients or outpatients at study sites (hospital and hospices in the United Kingdom).
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of oral symptoms (20) | 1 week
  Questionnaire

SECONDARY OUTCOMES:
Prevalence of physical / psychological symptoms | 1 week
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MD, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (11):
- United Kingdom (11):
  - Brighton & Sussex University Hospitals, Brighton, East Sussex
  - East Sussex Healthcare NHS Trust, Eastbourne, East Sussex
  - Pilgrims Hospice, Margate, Kent
  - Ellenor Lions Hospice, Northfleet, Kent
  - Hospice in the Weald, Pembury, Kent
  - Wisdom Hospice, Rochester, Kent
  - Frimley Park Hospital, Camberley, Surrey
  - Princess Alice Hospice, Esher, Surrey
  - Royal Surrey County Hospital, Guildford, Surrey
  - St. Wilfred's Hospice, Chichester, Wesr Sussex
  - St. Catherine's Hospice, Crawley, West Sussex

IPD SHARING:
Plan to Share IPD: No
Currently, there are no plans to make IPD available to other researchers

REFERENCES:
- [Result] Chang VT, Hwang SS, Feuerman M, Kasimis BS, Thaler HT. The memorial symptom assessment scale short form (MSAS-SF). Cancer. 2000 Sep 1;89(5):1162-71. doi: 10.1002/1097-0142(20000901)89:53.0.co;2-y. PMID 10964347
- [Derived] Davies A, Buchanan A, Todd J, Gregory A, Batsari KM. Oral symptoms in patients with advanced cancer: an observational study using a novel oral symptom assessment scale. Support Care Cancer. 2021 Aug;29(8):4357-4364. doi: 10.1007/s00520-020-05903-1. Epub 2021 Jan 8. PMID 33416995